CLINICAL TRIAL: NCT03724864
Title: Effect of a Daily Dose of Snacks Containing Mannitol or Stevia Rebaudiana as Sweeteners in High Caries Risk Schoolchildren
Brief Title: Edulcorants Effect in Caries Risk Schoolchildren
Acronym: STEVIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Guglielmo Campus, Associate Professor of Community Dentistry and Oral Epidemiology, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1138/L
Record Dates: First submitted 2018-10-25; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stevia snacks (Experimental): Children were instructed to use the snack twice a day, one in the morning and one in the afternoon during lesson breaks.
  Interventions: Dietary Supplement: delivery of snacks
- Maltitol snacks (Active Comparator): Children were instructed to use the snack twice a day, one in the morning and one in the afternoon during lesson breaks.
  Interventions: Dietary Supplement: delivery of snacks
- Sugared snacks (Placebo Comparator): Children were instructed to use the snack twice a day, one in the morning and one in the afternoon during lesson breaks.
  Interventions: Dietary Supplement: delivery of snacks

INTERVENTIONS:
Dietary Supplement: delivery of snacks — Subjects were randomly assigned to three groups (blue, green and yellow), receiving a single type of snack for 42 days. Block randomization ensured similar proportions of participants in each group. All subjects received snack packets (six cookies each) on a weekly basis. Children were instructed to use the snack twice a day, one in the morning and one in the afternoon during lesson breaks. Both participants and investigators were blinded to the treatment assignment.

SUMMARY:
This double-blind RCT aimed to evaluate the effect of sugar-free snacks on caries risk in 6-9 years-old schoolchildren. Considering a 20% difference among groups, the number of subjects needed per group was set in 87. Two-hundred-seventy-one children at risk for caries measured through Cariogram were selected and randomly assigned to three groups consuming twice a day snacks containing Stevia or Maltitol or sugar for 42 days. Parents filled out a standardized questionnaire regarding personal, medical and oral behavioural information. Bleeding on probing, plaque pH and cariogenic microflora were assessed at baseline (t0), after 21 (t1) and 42 days of snacks' use (t2) and 120 days after the end of use (t3). Cariogram was also repeated at t2.

ELIGIBILITY:
Inclusion Criteria:

* more than 1 initial carious lesion in the enamel (ICDAS 2-3),
* but no manifest lesion in the dentine,
* a salivary MS concentration ≥10^5 CFU/ml.

Exclusion Criteria:

* Subjects with a history of systemic diseases and antibiotic therapy within 30 days before baseline were excluded.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 271 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Caries risk reduction | 42 days
  calculation of the carie risk reduct using a standardised method aka "Cariogram"
reduction of salivary cariogenic bacteria | 42 days
  reduction of salivary cariogenic bacteria of one level eg from 1000000 to 10000 CFU/ml

SECONDARY OUTCOMES:
modification of the plaque-pH | 42 days
  reduction of the Area Under the Curve (AUC) at the critical level of pH of 6.2 and 5.7

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric dentistry dept, Sassari, Italy